CLINICAL TRIAL: NCT00609895
Title: The Incidence of Hypoglycemia in Insulin Glargine-Treated Subjects With Diabetes Mellitus Upon Switching Between Bedtime and Morning Dosing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4038
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine

INTERVENTIONS:
Drug: INSULIN GLARGINE

SUMMARY:
To compare the percentage of subjects with a glucose measurement < than or = to 56 mg/dL at any point of the 8-point glucose profiles during 3 consecutive days before vs. 3 consecutive days after switching insulin glargine dosing time from bedtime to morning and vs. 3 consecutive days after switching back to bedtime dosing of insulin glargine.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or type 2 diabetes mellitus diagnosis for at least 1 year Administration of insulin glargine for at least 2 months prior to screening; subjects must be on a stable dose of insulin glargine, + or - 15%, for at least 1 week prior to screening, given once daily at bedtime, and the dose must remain unchanged (+ or - 15%) during the screening period.
* If subjects are taking a short-acting insulin (e.g., regular human insulin, insulin lispro, or insulin aspart) or oral antidiabetic agents (e.g., a sulfonylurea, metformin, an alpha-glucosidase inhibitor, a thiazolidinedione, or a metiglinide), the subject must have been receiving these medications for at least 2 months prior to screening.
* For subjects taking an oral antidiabetic agent, the dose must be unchanged for the 2 weeks (4 weeks for a thiazolidinedione) prior to screening and should not be expected to be changed from the screening visit (day 14) through the final visit (day 11). The dose of any short-acting insulin may be changed if medically indicated.
* Males or non-pregnant females between the ages of 6 and 75 years; women must be postmenopausal for more than 2 years, surgically sterile, or agree to use a reliable contraceptive measure for the duration of the study. Reliable contraceptive measures include the following: systemic contraceptive (oral, implant, injections), diaphragm with intravaginal spermicide, cervical cap, intrauterine device, or condom with spermicide.
* Ability and willingness to perform blood glucose profiles using a plasma glucose meter provided at home over 11 consecutive days.
* HbA1c < than or = to 8.5% at screening.

Exclusion Criteria:

* Use of any other intermediate- or long-acting insulin (e.g., NPH, Ultralenter, Lenter) within the last 2 months prior to screening.
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol (e.g., systemic corticosteroids).
* History of hypoglycemia unawareness.
* Pregnancy (as determined by a serum pregnancy test at the screening visit).
* Breast-feeding.
* Treatment with any investigational drug in the 2 months prior to the screening visit.
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult.
* History of drug or alcohol abuse.
* Impaired hepatic function, as shown by but not limited to serum glutamic-oxaloacetic transaminase (SGPT, also known as alanine transaminase [ALT]) or serum glutamic-pyruvic transaminase (SGOT, also known as aspartate transaminase [AST]) above 2x the upper limit of normal range (ULN) measured at the screening visit.
* Impaired renal function, as shown by, but not limited to serum creatinine > than or = to 1.5 mg/dL (133 micromol/L) [males] or > than or = to1.4 mg/dL (124 micromol/L) [females] measured at the screening visit. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study. Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.
* Subjects who work the night shift.

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2004-01; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Compare % of subjects with glucose > or = to 56 mg/dL at any point of 8-point glucose profiles during 3 consecutive days | before vs. after switching dosing time from bedtime to morning and vs. after switching back to bedtime

SECONDARY OUTCOMES:
Compare % subjects with glucose measurements < or = to 72 mg/dL & < or = to 36 mg/dL at any point of the 8-point glucose profile during 3 consecutive days | before vs. after switching dosing time from bedtime to morning and vs. after switching back to bedtime
To compare the mean daily rate of hypoglycemia during 3 consecutive days | before vs. after switching dosing time from bedtime to morning and vs. after switching back to bedtime
To compare the changes from baseline in glucose values at each specific measurement time of the 8-point glucose profile during 3 consecutive days | before vs. after switching dosing time from bedtime to morning and vs. after switching back to bedtime
To compare the incidence of symptomatic hypoglycemia | at any time during 3 consecutive days before vs. after switching dosing time from bedtime to morning and vs. after switching back to bedtime
To evaluate overall safety and tolerability based on adverse event reporting, laboratory tests, and clinical examinations | at any time during the study

CONTACTS AND LOCATIONS:
Overall Officials: Judith Diaz, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Monterrey, Mexico